CLINICAL TRIAL: NCT00073775
Title: Epidemiology of Stress and the Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1239; R01HL072972 (NIH)
Record Dates: First submitted 2003-12-08; First posted 2003-12-10 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Hypertension; Hyperinsulinism; Insulin Resistance; Metabolic Syndrome X
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Hypertension; Hyperinsulinism; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, blood
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine the effects of psychological stress on the metabolic syndrome.

DETAILED DESCRIPTION:
BACKGROUND:

The metabolic syndrome identifies the clustering of lipid abnormalities, hypertension, hyperglycemia and abdominal obesity. It is a common and strong contributor to heart disease and diabetes and disproportionably affects older persons. Animal and small clinical studies have suggested that psychosocial stress is a risk factor for the metabolic syndrome. Underlying mechanisms may be through activation of the hypothalamopituitary-adrenal (HPA) axis causing hypercortisolemia, and, partly in turn, elevated inflammation and decreased sex hormone levels. However, longitudinal data showing that psychosocial stress indeed contributes to the onset and sequelae of the metabolic syndrome in the population at large, are lacking.

DESIGN NARRATIVE:

The primary objectives are to conduct data-analyses and biological sample analyses to examine the effect of psychosocial stress, as indicated by mood problems (depressive symptoms) and stressful social circumstances (poverty, negative life events, occupational stress, lack of emotional support), on the onset and sequelae of the metabolic syndrome. Secondary objectives are to examine underlying biological mechanisms in the effect of psychosocial stress on the metabolic syndrome. The investigators will use available data from two ongoing longitudinal community-based studies among older persons: the Health Aging and Body Composition (Health ABC) study (n=3,075, mean age=74 years, 52%=female, 42% African American) and the InChianti study (n=1,453, mean age=69 years, 56%=female). In both studies psychosocial stress and the metabolic syndrome are well defined, longitudinal data on sequelae (CVD events and diabetes onset) and onset of the metabolic syndrome are available, and potentially underlying biological variables were, or will be, assessed including 24-h urinary cortisol, serum sex steroid hormones (estradiol, testosterone, SHBG, DHEAS) and inflammatory markers (IL-6, IL-10, TNF-alpha, CRP, and various soluble cytokine receptors). The results of this study will help in designing future intervention trials that evaluate whether reducing stress and/or its physiological consequences, either by pharmacological treatment or behavioral intervention, could reduce incidence of the metabolic syndrome in the older general population.

ELIGIBILITY:
Age >70 years Community swelling

Ages: 70 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older persons
Sampling Method: Non-Probability Sample
Enrollment: 3075 (Actual)
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
There is no primary outcome | There is no time frame

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pahor, Principal Investigator — University of Florida